CLINICAL TRIAL: NCT03127059
Title: BEAT DB-study; Breathing Exercises in Asthma Targeting Dysfunctional Breathing-a Randomised Controlled Trial
Brief Title: Breathing Exercises in Asthma Targeting Dysfunctional Breathing
Acronym: BEAT_DB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Naestved Hospital (Other)
Collaborators: Zealand University Hospital (Other); Hvidovre University Hospital (Other); Aalborg University Hospital (Other); Bispebjerg Hospital (Other); TrygFonden, Denmark (Industry); Slagelse Hospital (Other); Region Zealand (Other); Association of Danish Physiotherapists (Other); Allergi og Lungeklinikken Helsingør (Unknown); Regionshospitalet Silkeborg (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Karen Hjerrild Andreasson, Ph.D.-Student, PT, Naestved Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJ-552
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Dysfunctional Breathing in Asthma
Keywords: Dysfunctional Breathing; Uncontrolled Asthma; Breathing Exercises; Adults
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Multi-centre, assessor-blinded, 2-arm randomised controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Three assessors (physiotherapists) will perform the objective assessment of capacity and lung parameters. Nurses in the outpatient departments will obtain data from medical records. The assessors and the nurses will be blinded for the allocation.
  The primary invenstigator will have no access to the data during the period of datacollection.
  Primary and most of the secondary outcomes will be patient-reported.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercises (Experimental): Individual instruction from a nurse at baseline aimed at knowledge on pharmacological treatment and optimized inhalation techniques. The participants will be encouraged to use online video instruction.
  Three physiotherapist-sessions of Breathing Exercises (BrEX) with duration of 60 minutes (the initial) and 30 minutes (other sessions) at week 1, 4, and 9. The participant is expected to do 10 minutes of home exercise twice daily. The entire intervention combines elements of the Papworth method, and the Buteyko technique.
  Interventions: Other: Breathing Exercises
- Usual care (Other): Individual instruction from a nurse at baseline aimed at knowledge on pharmacological treatment and optimized inhalation techniques. The participants will be encouraged to use online video instruction.
  Besides the individual instruction described above, patients will receive only short information given initially at recruitment. They are allowed to receive instruction in positive expiratory pressure-treatment and physiotherapy targeting other problems than dysfunctional breathing (DB).
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Breathing Exercises — Key points in the intervention are
  * Reduction (or normalising) of the respiration rate; use of rhythmic, nasal inspiration, diaphragmatic breathing; reduction of depth of breath, longer expiration; breath-holding at functional residual capacity.
  * Relaxation, especially the neck, jaw, tongue, and shoulders. Emphasizing the impact of gravity to the body.
  * Inclusion of the breathing modification into walking and other physical activities.
  * Daily home exercise of BrEX.
  Other Names: BrEX
  Arms: Breathing Exercises
Other: Usual care — Participants will receive only short information given initially at recruitment. No instruction or booklet will be distributed in the Usual care-Group.
  Other Names: UC
  Arms: Usual care

SUMMARY:
Dyspnoe can disable patients with asthma. Dysfunctional breathing (DB), resulting in dyspnoe, can mimic or exaggerate asthma. Around every forth patient with asthma have DB. Breathing exercises (BrEX) can improve asthma-related quality of live (QOL) in less severe asthma. No study has investigated the effect of BrEX on QOL neither on level of physical activity in severe asthma.

A randomised controlled multicentre trial will include 190 adults with poor asthma control (Asthma Control Questionnaire (ACQ6)-score≥0.8) from seven outpatient departments and one specialized private clinic. Patients will be allocated to either usual care (no intervention) or breathing exercises (BrEX)-treatment consisting of 12-week intervention including three physiotherapist-sessions focusing on breathing pattern modification (Papworth Method; Buteyko technique) in rest and activity and 10 minutes home-exercise twice daily. Primary outcome is change in Mini Asthma Quality of Life Questionnaire (MiniAQLQ) at six-months follow-up.

DETAILED DESCRIPTION:
In Denmark around 300,000 suffer from asthma. Dyspnoe can disable patients with asthma. Dysfunctional breathing (DB), resulting in dyspnoe, can mimic or exaggerate asthma. Around 20-29% of asthmatic patients have DB. Breathing exercises (BrEX) can improve asthma-related quality of life (QOL) and control of asthma symptoms in less severe asthma. No study has investigated the effect of BrEX on QOL neither on level of physical activity in severe asthma.

A randomised controlled multicentre trial will include 190 adults with poor asthma control (Asthma Control Questionnaire (ACQ6)-score≥0.8) from seven outpatient departments and one specialized private clinic. After optimizing of inhalation technique, patients will be allocated to either usual care (no intervention) or BrEX-treatment consisting of 12-week intervention including three physiotherapist-sessions focusing on breathing pattern modification (Papworth Method; Buteyko technique) in rest and activity and 10 minutes home-exercise twice daily. Primary outcome is change in Mini Asthma Quality of Life Questionnaire (MiniAQLQ) at six-months follow-up. Secondary outcomes are changes in ACQ6, Nijmegen Hyperventilation Questionnaire (NQ), Hospital Anxiety and Depression Scale (HAD), accelerometry (physical activity level, number of steps), 6 minutes walk distance, and forced expiratory volume in first second (FEV1), besides response of Global perceived effect rate (GPE) in asthma-related QOL and asthma control.

ELIGIBILITY:
Inclusion Criteria:

* Referred from GP to a secondary, out-patient respiratory clinic for lack of asthma control
* Pulmonologist-diagnosed asthma
* ≥ 2 consultations at a pulmonologist-lead asthma clinic
* ACQ6 ≥0.8
* Able to provide written informed consent.

Exclusion Criteria:

* Trained in breathing exercises by physiotherapist last 6 months
* Aged <18
* Pregnancy
* Not able to speak, read or understand Danish
* Any severe disease as judged by the responsible physician
* Participating in another pulmonary interventional research-project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2017-04-27 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Mini Asthma Quality of Life Questionnaire (MiniAQLQ) | Primary endpoint: Change from baseline to 6 months follow up. Secondary endpoints will be 3 and 12 months follow up.
  MiniAQLQ is a disease-specific patient-reported outcome on experiences during the previous two weeks. The original version of AQLQ (32 items) is recommended for clinical use, whereas this shortened version is suggested for research. In moderate to severe asthma cohorts, MiniAQLQ has good reliability (ICC 0.83-0.86) and strong validity (criteria validity to AQLQ, r≥0.80; construct validity against ACQ, r=0.69). MiniAQLQ has 15 items in four domains (symptoms, activity limitation, emotions, environment), which are answered using a 7-point Likert scale (1=maximum impairment; 7=no impairment).

SECONDARY OUTCOMES:
Asthma Control Questionnaire (ACQ6) | Change from baseline to 3, 6, and 12 months follow up
  Asthma Control Questionnaire (ACQ6) will be used in the 6 sub-score version omitting FEV1 % of predicted. The outcome-score is the mean of 6 sub-scores (5 questions about symptoms, 1 question in use of reliever medication (beta2-agonist)) using a 7-point Likert scale (0=fully controlled; 6=severely uncontrolled)
Nijmegen Questionnaire (NQ) | Change from baseline to 3, 6, and 12 months follow up
  A Nijmegen Questionnaire (NQ)-score > 23 suggests symptomatic hyperventilation, but is typically used to define DB.
Hospital Anxiety and Depression Scale (HAD) | Change from baseline to 3, 6, and 12 months follow up
  Hospital Anxiety and Depression Scale (HAD) uses a 0-21 scale; a low score indicates least mental health problems.
Global perceived effect rate (GPE) | At 3, 6, and 12 months follow up
  Global perceived effect rate (GPE) will be used as a retrospective evaluation of effect in asthma-related QOL as well as in asthma control on a 7-point Likert scale. GPE will only be measured at the follow ups.
Accelerometry (PAL, number of steps) | Change from baseline to 3 and 6 months follow up.
  Physical activity level (PAL) and numbers of steps will be measured by an accelerometer (BodyMedia SenseWear®) monitoring during 5 days
Spirometry (FEV1) | Change from baseline to 6 months follow up.
  Spirometry (MedikroPro) will be used to measure forced expiratory volume in first second in liter (FEV1).
6 Minutes Walk Distance (6MWD) | Change from baseline to 6 months follow up.
  6 Minutes Walk Distance (6MWD); 6MWD is the most typically used function-score in pulmonary research.

OTHER OUTCOMES:
Accelerometry (METs, TEE) | Change from baseline to 3 and 6 months follow up.
  Average metabolic equivalents (METs) and Total energy expenditure (TEE) will be measured by an accelerometer (BodyMedia SenseWear®) monitoring during 5 days.
Spirometry (FVC, PEF) | Change from baseline to 6 months follow up.
  Spirometry (MedikroPro) will be used to measure forced vital capacity (FVC), units liter, and peak expiratory flow rate (PEF), units liter/minute.
Inspiratory muscle strength (MIP) | Change from baseline to 6 months follow up.
  Inspiratory muscle strength (MIP), units cmH2O, will be measured by POWER Breathe®, KH2.
Adverse events (AE) | 12 months before baseline until 12 months follow-up.
  Adverse events (AE) e.g. emergency room visits will be extracted from medical report and from EasyTrial.Net (research database)
Register data from medical report | 12 months before baseline until 12 months follow-up.
  Comorbidity (types and numbers) and number of consultations at nurse and/or pulmonologist.
Register of Medical Product Statistics | 12 months before baseline until 12 months follow-up.
  For precise measure extraction of prescriptions on anti-asthmatic medication and comorbid medication on ATC-codes.
Foster Score | Change from inhalationcheck (before baseline) to 6 months follow up.
  Foster Score is used to investigate the number of days during the last seven days the participant took his/her asthma medication as prescribed. The participant is interviewed at the inhalationcheck, and will answer 0 to 7 referring to the number of days. Assessed again at 6 months follow up by questionnaire.
Adherence to physiotherapy-sessions | At 12 months follow-up.
  Adherence to the physiotherapist-sessions during the 12 weeks intervention will be investigated though data extracted in the electronically medical records.
Patient Acceptable Symptom State (PASS) | At 3, 6, and 12 months follow up.
  The dichotomous Patient Acceptable Symptom State (PASS) evaluates treatment success in the patient's perspective. The PASS will only be measured at the follow ups.
Participant-reported treatment failure. | At 3, 6, and 12 months follow up.
  If the participant answers 'no' to Patient Acceptable Symptom State (PASS) he/she will be asked to consider whether the treatment has failed.
Breath Holding Time (BHT) | Change from baseline to 6 months follow up.
  Time in seconds when nose is pinched at functional residual capasity until first respiratory muscle movement.
Count Scale (CS) | Change from baseline to 6 months follow up.
  Count Scale (CS) includes the count scale number (starting from 1 counting to as high as possible) and time spent while counting at a constant speed of 2 counts per second during one exhalation from max inspiratory level. CS has lower coefficient of variance at lower exercise level, than Borg Scale.
Borg CR10 | Change from baseline to 6 months follow up.
  Dyspnoe will be measured before and after 6MWD by the Borg CR10.
EuroQual-5Dimension (EQ-5D) | Change from baseline to 3, 6, and 12 months follow up.
  EuroQual-5Dimension (EQ-5D), a generic QOL tool that has high responsiveness, is translated into Danish and cross-cultural validated. EQ-5D index score of has been derived in the Danish population.
Socio Economic Status (SES) | Only assessed at baseline.
  Socio Economic Status (SES) includes education, work status, income.
Gender, Body Mass Index, smoking status, age | Only assessed at baseline.
  Participants gender, Body Mass Index (e.g., weight and height will be combined to report BMI in kg/m^2), smoking status (smoker/ former smoker/ non-smoker), and age will be self-reported at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Karen H Andreasson, PT MSc, Principal Investigator — University of Southern Denmark, Dep. of Physiotherapy and Occupational Therapy, Neastved-Slagelse-Ringsted Hospitals, Region Zealand, Denmark; Uffe Bødtger, MD PhD, Study Chair — University of Southern Denmark and Naestved Hospital; Søren T Skou, PT PhD, Study Chair — University of Southern Denmark and Naestved-Slagelse-Ringsted Hospitals; Mike Thomas, Prof MD PhD, Study Chair — University of Southampton and Aldermoor Health Centre, Southampton; Celeste Porsbjerg, Prof MD PhD, Study Chair — University of Copenhagen and Bispebjerg Hospital; Charlotte S Ulrik, Prof MD PhD, Study Chair — University of Copenhagen and Hvidovre Hospital; Peder G Fabricius, MD, Study Chair — Universityhospital Roskilde; Karin D Assing, MD, Study Chair — Aalborg University Hospital; Kirsten E Sidenius, MD PhD, Study Chair — Allergi og Lungeklinikken Helsingør; Charlotte Hyldgaard, MD, Study Chair — Diagnostisk Center, Regionshospitalet Silkeborg; Hanne Madsen, MD PhD, Study Chair — University of Southern Denmark and Odense University Hospital
Locations (8):
- Denmark (8):
  - Dep. of Physiotherapy and Dep. of Pulmonology, Silkeborg, Central Jutland
  - Dep. of Physiotherapy and Dep. of Pulmonology, Bispebjerg, Danish Capital Region
  - Allergi og Lungeklinikken Helsingør, Elsinore, Danish Capital Region
  - Dep. of Physiotherapy and Dep. of Pulmonology, Hvidovre, Danish Capital Region
  - Dep. of Physiotherapy and Dep. of Pulmonology, Aalborg, Region North
  - Dep. of Physiotherapy and Dep. of Pulmonology, Næstved, Region Sjælland
  - Dep. of Physiotherapy and Dep. of Pulmonology, Roskilde, Region Sjælland
  - Dep. of Physiotherapy and Dep. of Pulmonology, Odense, Region Syddanmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andreasson KH, Skou ST, Ulrik CS, Madsen H, Sidenius K, Jacobsen JS, Assing KD, Rasmussen KB, Porsbjerg C, Thomas M, Bodtger U. Protocol for a multicentre randomised controlled trial to investigate the effect on asthma-related quality of life from breathing retraining in patients with incomplete asthma control attending specialist care in Denmark. BMJ Open. 2019 Dec 31;9(12):e032984. doi: 10.1136/bmjopen-2019-032984. PMID 31892661
- [Result] Andreasson KH, Skou ST, Ulrik CS, Madsen H, Sidenius K, Assing KD, Porsbjerg C, Bloch-Nielsen J, Thomas M, Bodtger U. Breathing Exercises for Patients with Asthma in Specialist Care: A Multicenter Randomized Clinical Trial. Ann Am Thorac Soc. 2022 Sep;19(9):1498-1506. doi: 10.1513/AnnalsATS.202111-1228OC. PMID 35588357